CLINICAL TRIAL: NCT03597490
Title: Effectiveness of Multimodal Physical Therapy Combined With Exercise in Partial-thickness Rotator Cuff Tears: a Prospective Observational Study
Brief Title: Multimodal Physical Therapy With Exercise in Partial-thickness Rotator Cuff Tears
Status: Terminated | Type: Observational
Why Stopped: excessive dropout
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, ilker şengül, Principal Investigator, Izmir Katip Celebi University
Other Study IDs: 18.04.2018-150
Record Dates: First submitted 2018-07-02; First posted 2018-07-24 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Partial Thickness Rotator Cuff Tear
Keywords: Partial Thickness Rotator Cuff Tear; Physical Therapy
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Partial thickness rotator cuff tear: Patients with symptomatic non-traumatic partial thickness rotator cuff tear treated with multimodal physical therapy with exercise
  Interventions: Combination Product: Multimodal physical therapy with exercise

INTERVENTIONS:
Combination Product: Multimodal physical therapy with exercise — Multimodal physical therapy will compose of thermotherapy (hot pack or cold pack) and electrotherapy (transcutaneous electrical nerve stimulation or interferential current) and therapeutic ultrasound (at least two of them). Therapeutic exercise will compose of combination of range of motion, stretching, strengthening,neuromuscular and task specific exercises according to the clinical condition of patient under the supervision of a physiotherapist. Additionally, all patients will be allowed to carry on home exercise program.

SUMMARY:
The aim of this study is to investigate the early stage effectiveness of multimodal physical therapy with exercise in the conservative treatment of partial thickness rotator cuff tears.

DETAILED DESCRIPTION:
Although partial thickness rotator cuff tear prevalence is greater than those of full-thickness tear, most studies on conservative treatment are associated with full-thickness tears. In general, any physical therapy modality alone is not effective in the treatment of rotator cuff tears. It has been reported that multimodal physiotherapy may be more successful than monotherapy, but evidence in this regard is inadequate. Therefore this observational prospective study aiming to investigate the effectiveness of physiotherapy in the treatment of rotator cuff tears was planned. The null hypothesis of this study is that multimodal physical therapy combined with exercise has no effect on pain and function in the treatment of partial thickness rotator cuff tears. The alternative hypothesis is the opposite.

Patients will be assessed by standardized measures in terms of pain and function (American Shoulder and Elbow Surgeons standardized shoulder form: patient self report section), active range of motion (goniometric measurement) and quality of life (Western Ontario rotator cuff index) at baseline and first, third and 6th months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic partial thickness rotator cuff tear verified with magnetic resonance imaging or ultrasound imaging
* Prescription of multimodal physical therapy with exercise by a clinician other than investigators prior to inclusion in the study
* Covered by the social security system
* Giving informed consent to include in the study

Exclusion Criteria:

* Age of under 50
* Full thickness rotator cuff tear
* Radicular pain
* Glenohumeral osteoarthritis
* Calcific tendonitis
* Adhesive capsulitis
* History of physiotherapy in last 6 months
* Prior surgical treatment
* Contraindication to physical therapy and/or exercises

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic nontraumatic partial thickness rotator cuff tear
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-05-16 (Actual); Study Completion 2019-05-16 (Actual)

PRIMARY OUTCOMES:
Pain/function | Baseline to 6 months follow-up
  Pain and function are assessed by Turkish version of American Shoulder and Elbow Surgeons Standardized Shoulder Assessment Form, patient self-report section. It consists of two subscales including pain (one item) and function section (ten items). Pain and function subscales range between 0 and 50 with a maximum total score of 100. Lower pain subscale score means more pain, and lower function subscale score means more functional loss. The Turkish version of ASES standardized shoulder form:patient self reported section has been reported as reliable and valid.

SECONDARY OUTCOMES:
Disease specific health-related quality of life | Baseline to 6 months follow-up
  Disease specific health-related quality of life is assessed by Turkish version of Western Ontario Rotator Cuff Index.The Turkish version of the WORC index has been found a reliable and valid measurement tool. WORC index consists of 5 subscales including physical symptoms (6 items), sports and recreation (4 items), work (4 items), life style (4 items) and emotions (3 items). Each item is estimated based on 0-100 mm visual analogue scale. By summating the item scores, subscale scores and total scores are computed (possible total maximum score is 2100). Lower scores represents higher quality of life.

OTHER OUTCOMES:
Active range of motion of shoulder joint | Baseline to 6 months follow-up
  All active range of motion measurements of affected shoulder joint will be performed with a standard universal goniometer. While active range of motion of abduction and flexion (in degrees) will be measured in prone position, internal and external rotation measurement (in degrees) will be carried out in seating position while the shoulder is in 90 degrees abduction and elbow is in 90 degrees flexion.

CONTACTS AND LOCATIONS:
Overall Officials: ilker şengül, Principal Investigator — İzmir Katip Çelebi University
Locations (1):
- İlker Şengül, Izmir, In the USA Or Canada, Please Select..., Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Matthewson G, Beach CJ, Nelson AA, Woodmass JM, Ono Y, Boorman RS, Lo IK, Thornton GM. Partial Thickness Rotator Cuff Tears: Current Concepts. Adv Orthop. 2015;2015:458786. doi: 10.1155/2015/458786. Epub 2015 Jun 11. PMID 26171251
- [Background] Page MJ, Green S, McBain B, Surace SJ, Deitch J, Lyttle N, Mrocki MA, Buchbinder R. Manual therapy and exercise for rotator cuff disease. Cochrane Database Syst Rev. 2016 Jun 10;2016(6):CD012224. doi: 10.1002/14651858.CD012224. PMID 27283590
- [Background] Celik D, Atalar AC, Demirhan M, Dirican A. Translation, cultural adaptation, validity and reliability of the Turkish ASES questionnaire. Knee Surg Sports Traumatol Arthrosc. 2013 Sep;21(9):2184-9. doi: 10.1007/s00167-012-2183-3. Epub 2012 Aug 30. PMID 22932692
- [Background] El O, Bircan C, Gulbahar S, Demiral Y, Sahin E, Baydar M, Kizil R, Griffin S, Akalin E. The reliability and validity of the Turkish version of the Western Ontario Rotator Cuff Index. Rheumatol Int. 2006 Oct;26(12):1101-8. doi: 10.1007/s00296-006-0151-2. Epub 2006 Jun 24. PMID 16799776
- [Background] Kirkley A, Alvarez C, Griffin S. The development and evaluation of a disease-specific quality-of-life questionnaire for disorders of the rotator cuff: The Western Ontario Rotator Cuff Index. Clin J Sport Med. 2003 Mar;13(2):84-92. doi: 10.1097/00042752-200303000-00004. PMID 12629425
- [Background] Richards RR, An KN, Bigliani LU, Friedman RJ, Gartsman GM, Gristina AG, Iannotti JP, Mow VC, Sidles JA, Zuckerman JD. A standardized method for the assessment of shoulder function. J Shoulder Elbow Surg. 1994 Nov;3(6):347-52. doi: 10.1016/S1058-2746(09)80019-0. Epub 2009 Feb 13. PMID 22958838